CLINICAL TRIAL: NCT03231774
Title: Comparability of Hemodynamic Parameters Measured by Non-invasive Echocardiography and by Right Heart Catheterization
Status: Completed | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: HDZ-KA_011_HF
Record Dates: First submitted 2017-06-26; First posted 2017-07-27 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2018-09

CONDITIONS: Heart Failure
Keywords: Echocardiography; Right heart catheterization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to compare transthoracic Echocardiography TTE to the gold standard Right Heart Catheterization in Terms of accuracy to measure hemodynamic parameters.

DETAILED DESCRIPTION:
Chronic heart failure is a progressive disease in Western population. Echocardiography and right heart catheterization are important tools in the diagnosis and progress monitoring of heart failure.

Gold standard in diagnosis of hemodynamic parameters in patients with heart failure is right heart catheterization. However, this diagnostic device represents an invasive method that is additionally associated with high risks such as infections, vessel and nerve injuries. Echocardiography is probably in a position to determine hemodynamic parameters as reliably as right heart catheterization without additional health risk due to its non-invasive character. All procedures performed are part of clinical Routine. Patients do not undergo any study-specific procedure at all.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure NYHA I - IV

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for transthoracic echocardiography and right heart catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Measurement of systolic, diastolic and mean CVP | During a single right heart catheterization procedure
  CVP measured in mmHg

SECONDARY OUTCOMES:
Measurement of systolic, diastolic and mean PAP | During a single right heart catheterization procedure
  PAP measured in mmHg
Measurement of systolic, diastolic and mean RVP | During a single right heart catheterization procedure
  RVP measured in mmHg
Measurement of systolic, diastolic and mean PAWP | During a single right heart catheterization procedure
  PAWP measured in mmHg
Measurement of Cardiac Index CI | During a single right heart catheterization procedure
  CI measured in l/M/m²
Measurement of Cardiac Output CO | During a single right heart catheterization procedure
  CO measured in l/min
Transthoracic Echocardiography | During a single TTE examination
  Collected data will be analyzed for comparability

CONTACTS AND LOCATIONS:
Locations (1):
- Herz- und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fox H, Puehler T, Schulz U, Bitter T, Horstkotte D, Oldenburg O. Delayed recovery from Cheyne-Stokes respiration in heart failure after successful cardiac transplantation: a case report. Transplant Proc. 2014 Sep;46(7):2462-3. doi: 10.1016/j.transproceed.2014.06.063. PMID 25242802
- [Result] Szymczyk T, Sauzet O, Paluszkiewicz LJ, Costard-Jackle A, Potratz M, Rudolph V, Gummert JF, Fox H. Non-invasive assessment of central venous pressure in heart failure: a systematic prospective comparison of echocardiography and Swan-Ganz catheter. Int J Cardiovasc Imaging. 2020 Oct;36(10):1821-1829. doi: 10.1007/s10554-020-01889-3. Epub 2020 May 22. PMID 32445006